CLINICAL TRIAL: NCT06745388
Title: Evaluating the Impacts of Intravenous Magnesium Sulfate and Ketamine on Cramping Pain and Total Opioid Consumption Following Hysteroscopy: A Prospective, Randomized Trial
Brief Title: Magnesium and Cramping
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Roy Soto, MD, Staff physician, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-115
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Uterine Cramps; Postoperative Pain Management; Hysteroscopy
Keywords: hysteroscopy; magnesium sulfate; cramping; ketamine
MeSH Terms: conditions — Spasm | interventions — Magnesium Sulfate; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Magnesium, IV (Experimental): Intravenous magnesium 2 grams given over 20 minutes intra-operatively
  Interventions: Drug: Magnesium sulfate
- Ketamine, IV (Experimental): Intravenous ketamine 0.5 milligrams per kilogram dosed to ideal bodyweight, IV push intra-operatively
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): No administration of placebo infusion, ketamine or magnesium intra-operatively
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium sulfate — Receive intravenous magnesium intra-operatively
  Arms: Magnesium, IV
Drug: Ketamine — Receive IV push ketamine intra-operatively
  Arms: Ketamine, IV
Drug: Placebo — Receives no additional medication or infusion
  Arms: Placebo

SUMMARY:
Hysteroscopy (an exam to look inside the uterus) is one of the most frequently performed procedures for patients with cervical or uterine disorders. It is the gold standard for evaluating various intrauterine problems, pre-menopausal and post-menopausal abnormal uterine bleeding, as well as being a vital examination modality for infertility work-up. Although hysteroscopy is a minimally invasive procedure, it is still known to be a painful experience that requires effective analgesia (meaning pain reduction) to achieve maximum patient comfort and cooperation. Historically, opioids, particularly fentanyl, have held precedence as the primary agents for providing analgesia following surgery of this type. However, despite their efficacy, these agents come with notable drawbacks, including the potential for serious side effects such as respiratory depression, addiction, and postoperative nausea and vomiting.

Both magnesium and ketamine are routinely used to reduce pain following this procedure. Both drugs work on the N-methyl-D-aspartate (NMDA) receptor in the brain to reduce pain, and magnesium has an additional effect in that it can relax smooth muscles. Magnesium has been used successfully to reduce the pain associated with menstrual cramps, which is similar to the pain patients experience after hysteroscopy.

A recent study demonstrated the benefits of adding intravenous magnesium with routine anesthesia during hysteroscopy, revealing a significant decrease in postoperative pain and rescue analgesics. However, this study did not compare the effects of magnesium to ketamine, nor did they characterize the nature of the patients' pain. It is unclear if the pain reduction with magnesium comes from its effect on the NMDA receptor or from it's cramp-reduction effect. We seek to establish whether administering IV magnesium, compared to ketamine, can specifically mitigate uterine cramping pain and total opioid consumption in hopes of finding additional safe and effective pain modalities for patients.

This is a prospective, randomized trial enrolling participants undergoing an elective hysteroscopy or Dilation and Curettage (D&C) at Corewell Health William Beaumont University Hospital in Royal Oak. Participants will be randomized to 1 of 3 treatments: Intravenous (IV) Magnesium, IV Push Ketamine, or Placebo. Opioid consumption is recorded via the electronic medical record (EMR), while overall pain and cramping pain will be captured post-procedure in the hospital and 24 hours later via a phone call.

DETAILED DESCRIPTION:
This is a prospective, randomized trial enrolling participants undergoing an elective hysteroscopy or Dilation and Curettage (D&C) at Corewell Health William Beaumont University Hospital in Royal Oak. Participants will be initially contact via phone call 1 week prior to the procedure. If interested in participating, the study will be discussed pre-operatively and consent will be obtained. Baseline data including demographics, gynecological medical and surgical history, social history, allergies, current medications, ASA status, diagnosis, treatment and paucity will be collected.

The participant will be randomized to one of three study arms: IV magnesium, IV push ketamine, or placebo. The participants and evaluators will be blinded to the assigned study arm. The Principal Investigator and Anesthesiologist will not be blinded. All participants will receive standard of care anesthesia care and standard of care for the procedure.

Post-procedure, participants will receive standard of care pain management. Opioid consumption documented in the EMR will be recorded, and pain post-procedure pain will be assessed. Overall pain and cramping pain will be assessed using the Visual Analog Scale (VAS) at 1 hour, 2 hours, and 24 hours post procedure. The 24 hour pain assessment will be completed via phone.

Adverse events will be monitored for 24 hours post operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective hysteroscopy or dilation and curettage (D&C)
* American Society of Anesthesiologists (ASA) Physical Status 1 - 3
* Age 18 years or older

Exclusion Criteria:

* Chronic Pain Patients (taking opioids within one week of procedure)
* Psychiatric Disorders (current treatment for anxiety/depression)
* Allergies to any of the medications that will be administered
* Current use of magnesium, analgesics, antidepressants, anxiolytics, or opioids
* ASA Physical Status 4 or above
* Developmentally delayed patients that would not be able to verbalize pain scores
* Minors (under 18 years of age)
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Cramping Pain Following Hysteroscopy (1 hr post-operative) | 1 hour post-operatively
  Pain will be assessed 1 hour post-operatively using a Visual Analog Score (VAS). Pain is reported on a scale from 0-10; where 0=no cramping, and 10=cramping as bad as can be. A lower score indicates a better outcome.
Cramping Pain Following Hysteroscopy (2 hr post-operative) | 2 hours post-operatively
  Pain will be assessed 2 hours post-operatively using a Visual Analog Score (VAS). Pain is reported on a scale from 0-10; where 0=no cramping, and 10=cramping as bad as can be. A lower score indicates a better outcome.
Cramping Pain Following Hysteroscopy (24 hour post-operative) | 24 hours post-operatively
  Pain will be assessed 24 hours post-operatively using a Visual Analog Score (VAS). Pain is reported using a scale from 0-10; where 0=no cramping, and10=cramping as bad as can be. A lower score indicates a better outcome.
Overall Pain following hysteroscopy (1 hr post-operative) | 1 hour post-operatively
  Overall pain will be assessed 1 hour post-operatively using a 100-point Visual Analog Score (VAS). Pain is reported on a scale from 0-100; where 0=no pain, and 100=pain as bad as can be. A lower score indicates a better outcome.
Overall Pain following hysteroscopy (2 hr post-operative) | 2 hours post-operatively
  Overall pain will be assessed 2 hours post-operatively using a 100-point Visual Analog Score (VAS). Pain is reported on a scale from 0-100; where 0=no pain, and 100=pain as bad as can be. A lower score indicates a better outcome.
Overall Pain following hysteroscopy (24 hr post-operative) | 24 hours post-operatively
  Overall pain will be assessed 24 hours post-operatively using a 100-point Visual Analog Score (VAS). Pain is reported on a scale from 0-100; where 0=no pain, and 100=pain as bad as can be. A lower score indicates a better outcome.

SECONDARY OUTCOMES:
Opioid consumption Following Hysteroscopy | 24 hours post-operatively
  Opioid consumption will be recorded in morphine milligram equivalents (MME). The total MME for all patients for each intervention arm. A lower number indicates a better outcome as fewer opioids were consumed for pain management post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ray Soto, MD, Principal Investigator — Corewell Health East
Locations (1):
- Corewell Health William Beaumont University Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual patient data (IPD) may be made available on request to the principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: Available following final closure of study and publication of results (anticipated December 2026) for up to 2 years (anticipated December 2028).
Access Criteria: Deidentified data may be made available on request to the principal investigator for legitimate research use.